CLINICAL TRIAL: NCT06796712
Title: BiomeBakery: A Randomised Controlled Parallel Trial to Investigate the Cognitive, Affective, Inflammatory and Metabolic Effects of Chronic Prebiotic-fortified Functional Bakery Product Intervention in Older Adults
Brief Title: BiomeBakery Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Innovate UK (Other Government); Biotechnology and Biological Sciences Research Council (Other); Myota Limited (Unknown); Puratos Limited (Unknown); Thriva Limited (Unknown)
Responsible Party: Principal Investigator, Piril Hepsomali, Principle Investigator, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UREC 24/36
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cognition; Affect (Mental Function); C Reactive Protein
Keywords: prebiotics; fibre; cognition; depression; anxiety; inflammation
MeSH Terms: conditions — Depression; Anxiety Disorders; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active: Prebiotic fibre-fortified bread roll (Experimental): Subjects will consume a prebiotic fibre-fortified bread roll (10g of added prebiotic fibre/day).
  Interventions: Dietary Supplement: Prebiotic fibre fortified bread roll
- Placebo: Regular bread roll (Placebo Comparator): Subjects will consume a regular bread roll (0g of added prebiotic fibre blend/day).
  Interventions: Dietary Supplement: Regular bread roll

INTERVENTIONS:
Dietary Supplement: Prebiotic fibre fortified bread roll — Subjects will consume a prebiotic fibre-fortified bread roll (10g of added prebiotic fibre/day).
  Arms: Active: Prebiotic fibre-fortified bread roll
Dietary Supplement: Regular bread roll — Subjects will consume a regular bread roll (0g of added prebiotic fibre blend/day).
  Arms: Placebo: Regular bread roll

SUMMARY:
This study aims to investigate the chronic effects of prebiotic fibre-fortified functional bakery product on cognitive, affective, inflammatory, metabolic, and anthropometric outcomes in healthy adults aged 60-75 years with mild to moderate subjective cognitive complaints.

DETAILED DESCRIPTION:
This study will employ a double-blind, randomised, placebo-controlled parallel design to investigate the chronic effects of an 12 week prebiotic fibre-fortified functional bakery product on cognitive, affective, inflammatory, metabolic, and anthropometric outcomes in healthy older adults with mild to moderate subjective cognitive complaints.

Seventy four participants will be randomised (1:1 ratio, matched by age, sex, and fibre intake) to Intervention or Placebo groups where they will be consuming a prebiotic fibre-fortified functional bakery product (containing 10g prebiotic fibre/day) or a regular bakery product (containing 0g prebiotic fibre/day), respectively, for 12-weeks. Outcome measures will be acquired before and after a 12-week chronic supplementation. These will include cognitive measures of overall cognitive functioning, immediate and delayed verbal memory, executive functions; affective measures of depression and anxiety symptomatology; gastrointestinal symptomatology; inflammatory measure of high sensitivity C-reactive protein (hs-CRP); metabolic measures of lipid profiles (total-C, LDL-C, HDL-C, triglycerides), Hemoglobin A1c (HbA1c) and systolic and diastolic blood pressure; and anthropometric measures of height, weight, hip and waist circumference.

ELIGIBILITY:
Inclusion Criteria:

* Aging between 60-75 years old
* Having normal vision and hearing
* Having a normal body mass index (BMI<30)
* Having mild to moderate subjective cognitive complaints
* Consuming bread (5 or more times a week)

Exclusion Criteria:

* Smoking
* Having food allergies
* Following restrictive and/or unbalanced diets
* Changing dietary intake majorly in past month
* Being diagnosed with any psychiatric or neurologic conditions (e.g. schizophrenia, depression, dementia) including eating disorders
* Being diagnosed with any cardiometabolic diseases (including type II diabetes and cardiovascular disease), or suffering from hypertension or thrombosis related disorders or suffer from thyroid disease
* Being anaemic
* Currently taking anticoagulants, antiplatelet medication, antidepressants, proton-pump inhibitors
* Currently consuming prebiotic or probiotic supplements
* Continuous antibiotic use for > 3 days within 1 month prior to enrolment
* Continuous use of weight-loss drug for > 1 month before screening
* Having a significant gastrointestinal (GI) condition affecting absorption including (but not limited to) inflammatory bowel disease; total colectomy or bariatric surgery; irritable bowel disease; end stage renal disease; active cancer, or treatment for any cancer, in last 3 years
* Having a high fibre intake defined as > 20g of fibre/day
* Wheat and/or gluten intolerance and having coeliac disease

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment score | From baseline (pre intervention) to week 12 (post intervention)
  Composite measure of global cognitive function - the total possible score is 30 points; a score of 26 or above is considered normal.
hs-CRP levels | From baseline (pre intervention) to week 12 (post intervention)
  High- sensitivity C-Reactive protein (hs-CRP) levels in plasma samples

SECONDARY OUTCOMES:
Immediate Word Recall from the Rey Auditory Verbal Learning Task | From baseline (pre intervention) to week 12 (post intervention)
  Participants will be presented with a sequential list of 15 words, at a rate of 1 word per second. The participant will then have 60s to say out loud as many of these words as possible, with the resulting score recorded as a percentage of accuracy.
Delayed Word Recall from the Rey Auditory Verbal Learning Task | From baseline (pre intervention) to week 12 (post intervention)
  After a period of time subject are asked to recall as many words as possible from list A
Word Recognition from the Rey Auditory Verbal Learning Task | From baseline (pre intervention) to week 12 (post intervention)
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
EPIC Norfolk Food Frequency Questionnaire (FFQ) | From baseline (pre intervention) to week 12 (post intervention)
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.
Working Memory Questionnaire Score | From baseline (pre intervention) to week 12 (post intervention)
  A measure assessing short-term storage, attention, and executive control
Gastrointestinal Symptom Rating Scale Scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of gastrointestinal symptoms that includes 15-items (combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation) .
Geriatric Depression Scale scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of depression that includes 15-items.
Geriatric Anxiety Inventory scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of anxiety that includes 20-items.
Positive and Negative Affect Schedule (PANAS) | From baseline (pre intervention) to week 12 (post intervention)
  A 20-item questionnaire measuring positive and negative affect.
Lipid profiles | From baseline (pre intervention) to week 12 (post intervention)
  Total-Cholesterol, Low-density lipoprotein cholesterol (LDL-C), High-density lipoprotein cholesterol (HDL-C), and triglycerides will be assessed.
Hemoglobin A1c (HbA1c) | From baseline (pre intervention) to week 12 (post intervention)
  Hemoglobin A1c (HbA1c) will be assessed.
Blood Pressure | From baseline (pre intervention) to week 12 (post intervention)
  Systolic and diastolic blood pressure (in mmHg) will be measured.
Anthropometric outcomes | From baseline (pre intervention) to week 12 (post intervention)
  Hip and waist circumference (in cm) will be measured. Additionally, weight (in kg) and height (in m) will be combined to report BMI in kg/m^2.

OTHER OUTCOMES:
FiberScreen Scores | Baseline (pre intervention)
  A questionnaire that assesses fibre intake. It will be used to screen participants. Individuals who adhere to a high fibre diet (>20g fibre/day) will be excluded from the study.
Telephone Interview for Cognitive Status-40 | Baseline (pre intervention)
  A questionnaire that assesses cognitive status. It will be used to screen participants. Only individuals who score between 6 and 20 (depicting mild to moderate subjective cognitive complaints) will be included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, School of Psychology and Clinical Languages, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No